CLINICAL TRIAL: NCT03804151
Title: The Impact of the FitSpirit Physical Activity Approach on Different Health Parameters of Canadian Adolescent Girls: the Protocol of a Large, Longitudinal Quasi-experimental Study
Brief Title: Long-term Evaluation of the FitSpirit Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: FitSpirit (Unknown); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Marie-Ève Mathieu, Associate professor, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FitSpirit Evaluation LAPS
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Sedentary Behavior
Keywords: Exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FitSpirit Intervention (Experimental): FitSpirit physical activities and events are organized by participants' schools during the school year. Girl-only activities such as physical activity sessions, speaking engagements, turnkey running program and special events can be offered. The number, type and frequency of activities are decided by each school.
  Interventions: Behavioral: FitSpirit intervention

INTERVENTIONS:
Behavioral: FitSpirit intervention — The study evaluates the effects of the FitSpirit intervention on divers health markers of adolescents. Participants freely register to the intervention via their school. Physical activities and event are organized by the schools with the help of the FitSpirit organization.

SUMMARY:
This study evaluates the long-term effects of the FitSpirit extra-curricular, girl-only intervention on numerous health outcomes of adolescent girls.

ELIGIBILITY:
Inclusion Criteria:

* Attend high-school registered to FitSpirit

Exclusion Criteria:

-

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participants who self-identify as female adolescents are eligible to the intervention.
Enrollment: 1200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity participation | Markers re evaluated at the beginning and the end of each school years (approximately 7 months appart)
  An online questionnaire assesses physical activity participation. It is measured using the number of days per week the participant are active more than 60 min/day (scale 0 to 7 days/week).
Eating habits | Markers re evaluated at the beginning and the end of each school years (approximately 7 months appart)
  An online questionnaire assesses eating habits. They are measured using the number of servings consumed per week for each of the different food categories (fruits, vegetables, juice, milk products, sweetened beverages, and fast food). No aggregation is done.
Sleep habits | Markers re evaluated at the beginning and the end of each school years (approximately 7 months appart)
  An online questionnaire assesses sleep habits. They are evaluated based on the usual number of hours of sleep (hours per night).
Physical self-efficacy | Markers re evaluated at the beginning and the end of each school years (approximately 7 months appart)
  Physical self-efficacy is assessed using an online questionnaire by asking the participants their level of agreement with 12 statements, using a 5 level scale. Points are attributed to each answer (Disagree totally: 1; Somewhat disagree: 2; Neutral: 3; Somewhat agree: 4; Agree totally: 5). Total score is used to compare the participants and highest score represents a better outcome.
Physical self-perception | Markers re evaluated at the beginning and the end of each school years (approximately 7 months appart)
  Physical self-perception is evaluated using an online questionnaire presenting 2 sets of 7 silhouettes. Participants identify first the silhouette representing best their current body image. They then identify the silhouette representing their desired body image (slimmest silhouette: 1 point; fattest silhouette: 7 points). Satisfaction of body image is calculated by the difference between the 2 answers. Smaller difference score represent better satisfaction of body image.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eve Mathieu, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The database, excluding individual information, will be shared with the co-investigators of the study.

REFERENCES:
- [Derived] Leduc G, Gilbert JA, Ayotte A, Moreau N, Drapeau V, Lemoyne J, Monthuy-Blanc J, Tremblay J, Mathieu ME. The FitSpirit approach for increasing physical activity in canadian teenage girls: protocol of a longitudinal, quasi-experimental study. BMC Public Health. 2021 Jan 28;21(1):229. doi: 10.1186/s12889-021-10200-5. PMID 33509155